CLINICAL TRIAL: NCT04561362
Title: Phase I/II Study of the Safety, Pharmacokinetics, and Preliminary Clinical Activity of BT8009 in Patients With Nectin-4 Expressing Advanced Malignancies
Brief Title: Study BT8009-100 in Subjects With Nectin-4 Expressing Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BicycleTx Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT8009-100
Record Dates: First submitted 2020-09-14; First posted 2020-09-23 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Urinary Bladder Neoplasm; Triple Negative Breast Neoplasms; Hormone Receptor Positive, HER2-negative Neoplasms; Hormone Receptor Positive, HER2-low Neoplasms; Breast Neoplasms; Non-Small-Cell Lung Neoplasms; Ovarian Neoplasm; Advanced Solid Tumor
Keywords: Nectin-4; Solid tumor; Transitional urothelial carcinoma; Renal insufficiency
MeSH Terms: conditions — Urinary Bladder Neoplasms; Triple Negative Breast Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Renal Insufficiency | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A-1 -BT8009 Monotherapy Dose Escalation (Experimental): Participants will receive escalating doses of BT8009.
  Interventions: Drug: BT8009
- Part A-2 -BT8009 in Combination with Pembrolizumab Dose De-Escalation (Experimental): Participants will receive BT8009 and a standard dose of pembrolizumab.
  Interventions: Drug: BT8009; Drug: Pembrolizumab
- Cohort B-1 - BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Cohort B-2- BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Cohort B-3- BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009. .
  Interventions: Drug: BT8009
- Cohort B-4- BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Cohort B-5- BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Cohort B-6- BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Cohort B-7- BT8009 in Combination with Pembrolizumab Dose Expansion (Experimental): Participants will receive a selected dose of BT8009 and standard dose of pembrolizumab.
  Interventions: Drug: BT8009; Drug: Pembrolizumab
- Part C - Renal Insufficiency BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Part D - BT8009 Monotherapy Supplementary PK (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Part B-8 - BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009
- Part B-9 - BT8009 Monotherapy Dose Expansion (Experimental): Participants will receive a selected dose of BT8009.
  Interventions: Drug: BT8009

INTERVENTIONS:
Drug: BT8009 — Bicyclic Toxin Conjugate (BTC) administered either weekly (i.e., on Days 1, 8, 15, and 22) or biweekly (Days 1 and 15) on a 28-day cycle or on Days 1 and 8 of a 21-day cycle for participants in A-1. Participants in Cohorts A-2 and B-7 will receive BT8009 weekly on 21-day cycle. Participants in Parts B-1-B-6 will receive BT8009 weekly either on a 21-day or 28-day cycle. Participants in Parts B-8 and B-9 will receive BT8009 on Days 1 and 8 of a 21-day cycle. Participants in Cohort C will receive BT8009 once weekly (i.e., on Days 1, 8, 15, and 22) on a 28-day cycle. Participants in Part D will receive BT8009 once weekly on a 28-day cycle.
Drug: Pembrolizumab — Participants in Cohorts A-2 and B-7 will receive 200 mg IV over 30-minute infusion of pembrolizumab on Day 1 of each Q3W.
  Other Names: Keytruda
  Arms: Cohort B-7- BT8009 in Combination with Pembrolizumab Dose Expansion; Part A-2 -BT8009 in Combination with Pembrolizumab Dose De-Escalation

SUMMARY:
This study is a Phase I/II, multicenter, first-in-human, open-label dose-escalation study of BT8009 given as a single agent and in combination with pembrolizumab in participants with advanced solid tumors associated with Nectin-4 expression or in participants with advanced solid tumor malignancies having renal insufficiency. The primary endpoints are: Dose limiting toxicities (Parts A-1 and A-2), Overall response rate per RECIST v1.1 (Parts B1-B7), Safety and tolerability (Parts B-8, B-9 and C), and characterization of the pharmacokinetics (Part D).

DETAILED DESCRIPTION:
This study will assess the safety and tolerability of BT8009 alone and in combination with pembrolizumab in patients with select advanced solid tumors. BT8009 will be given as a single agent in 3 different dosing schedules- weekly (28 day cycle), biweekly (28 day cycle) or dosing on day 1 and day 8 of a 3-weekly (21 day cycle) and in combination with pembrolizumab. There are four parts to this study. Part A is a dose escalation in patients with select advanced solid tumors primarily designed to evaluate safety and tolerability of BT8009 as monotherapy or in combination with pembrolizumab and to determine a recommended Phase II dose (RP2D). Following a selection of an RP2D, Part B, a dose expansion portion, will be initiated with the primary objective of clinical activity of BT8009 as a monotherapy or in combination with pembrolizumab in patients with select advanced solid tumors. Additionally Parts B-8 and B-9 will evaluate the safety and tolerability of an alternate dose and schedule of BT8009 monotherapy. Part C will evaluate safety and tolerability of RP2D in patients with renal insufficiency. Part D will further characterize the pharmacokinetics of BT8009 and MMAE.

ELIGIBILITY:
Key Inclusion Criteria

* Life expectancy ≥12 weeks.
* Patients must have measurable disease per RECIST 1.1.
* Part A-1 cohorts:
* Must have exhausted all standard treatment options, including appropriate targeted therapies; or patients for which no standard therapy is considered appropriate
* Patients with advanced, histologically confirmed urothelial (transitional cell) carcinoma that recurred after or has been refractory to prior therapy (fresh tumor biopsy or an archived sample must be submitted); or
* Patients with advanced, histologically confirmed pancreatic, breast, non-small-cell lung cancer (NSCLC), gastric, esophageal, head and neck, or ovarian tumors that recurred after or has been refractory to prior therapy (fresh tumor biopsy or an archived sample testing for Nectin-4 expression).
* Part A-2:
* Must have exhausted all standard treatment options, including appropriate targeted therapies; or patients for which no standard therapy is considered appropriate
* Patients with advanced, histologically confirmed urothelial (transitional cell) carcinoma that have progressed following prior therapy
* Cohort B-1: Histologically documented urothelial carcinoma, previously treated with enfortumab vedotin (EV). Patients with resectable, locally advanced urothelial carcinoma are ineligible. Must have had progression or recurrence of urothelial cancer during or following receipt of most recent therapy.
* Cohort B-2 and B-3: Histologically documented urothelial carcinoma, not previously treated with enfortumab vedotin (EV). Patients with resectable, locally advanced urothelial carcinoma are ineligible. Must have had progression or recurrence of urothelial cancer during or following receipt of most recent therapy.
* Cohort B-4: Patients with histologically confirmed non-mucinous epithelial ovarian, fallopian tube, or primary peritoneal cancer that is Stage III or IV according to the International Federation of Gynecology and Obstetrics (FIGO) or tumor, node and metastasis staging criteria that have progressed following prior therapy.
* Cohort B-5: Patients with triple-negative breast cancer confirmed negative for estrogen receptor (ER) and progesterone receptor (PR) and negative for human epidermal growth factor receptor 2 (HER2) (i.e., triple-negative) that have progressed following prior therapy.
* Cohort B-6: Patients with histologically confirmed non-small cell lung cancer (NSCLC) with no actionable mutations, such as Epidermal Growth Factor Receptor (EGFR) mutation, anaplastic lymphoma kinase (ALK) fusion oncogene, or ROS1 that have progressed following prior therapy.
* Cohort B-7: Locally advanced or metastatic, histologically confirmed urothelial (transitional cell) carcinoma, ineligible for cisplatin, no prior systemic anticancer treatment for advanced urothelial carcinoma.
* Cohort B-8: Locally advanced (unresectable) or metastatic, histologically confirmed breast cancer, either TNBC or hormone receptor (HR) positive and HER-2 negative according to ASCO/CAP guidelines and up to 3 prior lines of therapy for advanced (unresectable) or metastatic disease.
* Cohort B-9: Histologically confirmed advanced/metastatic squamous or non-squamous NSCLC, negative for oncogenic driver mutations (EGFR, KRAS, ALK, BRAF, MET, ERRB2).
* Cohort C renal insufficiency cohort: Patients with histologically documented urothelial carcinoma, ovarian, triple negative breast, or non-small cell lung cancer that have been previously treated with a locally approved therapy.
* Part D supplementary PK: Patients must have histologically confirmed urothelial (transitional cell) carcinoma (patients with squamous differentiation or mixed cell types are eligible); ovarian; triple-negative breast; or non-small cell lung cancer that have been previously treated with a locally approved therapy.

Key Exclusion Criteria (all patients):

* Clinically relevant troponin elevation
* Uncontrolled diabetes
* Known active or untreated CNS and/or carcinomatous meningitis
* Grade ≥2 peripheral neuropathy
* Active keratitis or corneal ulcerations
* Patients with uncontrolled hypertension
* History of another malignancy within 3 years before first dose of BT8009 or residual disease from a previously diagnosed malignancy (with some exceptions).
* Active systemic infection requiring therapy, or fever within the last 14 days prior to first dose of BT8009.
* Prior Stevens-Johnson syndrome/toxic epidermal necrolysis on any MMAE-conjugated drug
* Parts A-2 and B-7 Pembrolizumab Combination Cohorts:
* Prior organ transplant (including allogeneic)
* Diagnosis of clinically relevant immunodeficiency
* History of interstitial lung disease
* Parts B-2 and B-3: Prior treatment with enfortumab vedotin Other protocol-defined Inclusion/Exclusion criteria may apply
* Parts B-8 and B-9: Prior treatment with an ADC containing an MMAE (vedotin) payload.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Parts A-1, A-2 and C: Number of participants with treatment emergent adverse events, receiving BT8009 as a monotherapy or in combination with pembrolizumab to assess safety and tolerability. | From cycle 1 day 1 until 30 days after the end of treatment or approximately 1 year
  Safety reported as incidence of treatment-emergent adverse events using CTCAE v5.0 criteria.
Parts A-1 and A-2 (escalations): Number of participants with dose limiting toxicities on BT8009 as a monotherapy or in combination with pembrolizumab | 28 days (for cycles that are either 21 or 28 days in length depending on dosing schedule assigned)
  Number of patients who experience dose limiting toxicities BT8009 when given as a monotherapy or in combination with pembrolizumab.
Part B1-B7: Objective response rate (ORR) to assess the clinical activity of BT8009 as a monotherapy or in combination with pembrolizumab using RECIST 1.1. | Every 8 weeks for 12 months then every 12 weeks thereafter until disease progression or, death, or up to three years
  Proportion of participants with confirmed complete response or partial response to BT8009 as a monotherapy or in combination with pembrolizumab according to RECIST 1.1 criteria.
Part D: Maximum plasma concentration (Cmax) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment or for up to 1 year
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone.
Part D: Minimum plasma concentration (Cmin) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment or for up to 1 year
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone
Part D: Area under the plasma concentration-time curve (AUC) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment or for up to 1 year
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone.
Part D: Elimination half-life (t1/2) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment or for up to 1 year
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone.
PartsB-8, B-9: Number of participants with treatment emergent adverse events receiving an alternative dosing regimen of BT8009 monotherapy to assess safety and tolerability. | From cycle 1 day 1 until at least 30 days after the end of treatment (each cycle is 21 days)
  Number of participants with advanced solid tumor malignancies associated with Nectin-4 expression receiving an alternative dose regimen of BT8009 as a monotherapy who experience treatment-emergent adverse events using CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Parts B-1-B-7: Number of participants with treatment emergent adverse events receiving BT8009 as a monotherapy or in combination with pembrolizumab to assess safety and tolerability. | From cycle 1 day 1 until at least 30 days after the end of treatment (each cycle is 21 or 28 days depending on the assigned dosing schedule)
  Number of participants with advanced solid tumor malignancies associated with Nectin-4 expression receiving BT8009 as a monotherapy or in combination with pembrolizumab who experience treatment-emergent adverse events using CTCAE v5.0 criteria.
Part B: Duration of Response time to assess preliminary anti-tumor activity of BT8009 as a monotherapy or in combination with pembrolizumab | Every 8 weeks for 12 months then every 12 weeks thereafter until disease progression or, death, or up to three years
  Duration of objective response (complete or partial response) by RECIST 1.1 in participants receiving BT8009 as a monotherapy or in combination with pembrolizumab
Part B: Clinical benefit rate to assess the clinical activity of BT8009 as a monotherapy or in combination with pembrolizumab | Every 8 weeks Parts A-1, A-2, and C) and every 9 weeks (cohorts B-8 and B-9) for 12 months then every 12 weeks thereafter until disease progression or death or up to 3 years
  Proportion of participants who have complete response (CR), partial response (PR), or stable disease (SD) for at least 16 weeks according to RECIST Version 1.1 criteria.
Part B: Progression-free survival time to assess the clinical activity of BT8009 as a monotherapy or in combination with pembrolizumab. | Every 8 weeks for the first 12 months then every 12 weeks until disease progression or death for up to three years
  The time from the first day of study drug administration (Day 1) to disease progression according to RECIST 1.1 criteria in participants receiving BT8009 as a monotherapy or in combination with pembrolizumab.
Part B: Overall survival time to assess the clinical activity of BT8009 as a monotherapy or in combination with pembrolizumab using RECIST 1.1 | Every 8 weeks for the first 12 months then every 12 weeks until death, then every 3 months for up to 1 year after last patient accrued
  The time from start of study drug administration (Day 1) until death due to any cause in participants receiving BT8009 as a monotherapy or in combination with pembrolizumab.
Cohorts B-4, B-5, and B-6: Objective response rate by Nectin-4 status of BT8009 as a monotherapy in patients with selected solid tumor using RECIST 1.1. | Every 8 weeks for the first 12 months then every 12 weeks until disease progression or death for up to three years
  Proportion of participants with confirmed complete response or partial response to BT8009 as a monotherapy according to RECIST 1.1 criteria categorized by Nectin-4 expression status.
Parts A-1, A-2, B-8, B-9, and C: Objective response rate to assess preliminary anti-tumor activity of BT8009 as a monotherapy or in combination with pembrolizumab. | Every 8 weeks for the first 12 months then every 12 weeks until disease progression or death or up to three years
  Proportion of participants with advanced solid tumor malignancies associated with Nectin-4 expression or advanced solid tumor malignancies having renal insufficiency with confirmed complete response or partial response according to RECIST 1.1 criteria
Parts A-1, A-2, C and D: Duration of Response time to assess preliminary anti-tumor activity of BT8009 as a monotherapy or in combination with pembrolizumab. | Every 8 weeks for the first 12 months then every 12 weeks until disease progression or death or up to three years
  Duration of objective response (complete or partial response) by RECIST 1.1 in participants with advanced solid tumor malignancies associated with Nectin-4 expression or advanced solid tumor malignancies having renal insufficiency receiving BT8009 as a monotherapy or in combination with pembrolizumab.
Parts A-1, A-2, C and D: Clinical benefit rate to assess preliminary anti-tumor activity of BT8009 as a monotherapy or in combination with pembrolizumab | Every 8 weeks for the first 12 months then every 12 weeks until disease progression for up to 3 years
  Proportion of participants with advanced solid tumor malignancies associated with Nectin-4 expression or advanced solid tumor malignancies having renal insufficiency who have complete response (CR), partial response (PR) or stable disease (SD) for at least 16 weeks according to the RECIST Version 1.1 criteria.
Parts A-1, A-2, C and D: Progression-free survival time (months) to assess preliminary anti-tumor activity of BT8009 as a monotherapy or in combination with pembrolizumab | Every 8 weeks for the first 12 months then every 12 weeks until disease progression or death for up to three years
  The time from start of study drug administration until disease progression according to RECIST 1.1 in participants with advanced solid tumor malignancies associated with Nectin-4 expression or advanced solid tumor malignancies having renal insufficiency receiving BT8009 as a monotherapy or in combination with pembrolizumab.
Parts A-1, A-2, C and D: Overall survival time (months) to assess preliminary anti-tumor activity of BT8009 as a monotherapy or in combination with pembrolizumab. | Every 8 weeks for the first 12 months then every 12 weeks until disease progression, then every 3 months for up to 1 year after last patient is accrued
  The time from start of study drug administration until death due to any cause in participants with advanced solid tumor malignancies associated with Nectin-4 expression or advanced solid tumor malignancies having renal insufficiency receiving BT8009 as a monotherapy or in combination with pembrolizumab.
Part A, B and C: Maximum plasma concentration (Cmax) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy and in combination with pembrolizumab. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone and in combination with pembrolizumab.
Part A, B and C: Minimum plasma concentration (Cmin) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy and in combination with pembrolizumab. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone and in combination with pembrolizumab.
Part A, B and C: Area under the plasma concentration-time curve (AUC) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy and in combination with pembrolizumab. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone and in combination with pembrolizumab.
Part A, B and C: Elimination half-life (t1/2) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy and in combination with pembrolizumab. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations of BT8009 and MMAE from all participants taking BT8009 alone and in combination with pembrolizumab.
Part C: Maximum plasma concentration (Cmax) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations (for impact of renal impairment) of BT8009 and MMAE from Part C participants taking BT8009 as a monotherapy.
Part C: Minimum plasma concentration (Cmin) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherap. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations (for impact of renal impairment) of BT8009 and MMAE from Part C participants taking BT8009 as a monotherapy.
Part C: Area under the plasma concentration-time curve (AUC) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations (for impact of renal impairment) of BT8009 and MMAE from Part C participants taking BT8009 as a monotherapy.
Part C: Elimination half-life (t1/2) of BT8009 and monomethyl auristatin E (MMAE) when given as monotherapy. | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Plasma concentrations (for impact of renal impairment) of BT8009 and MMAE from Part C participants taking BT8009 as a monotherapy.
All cohorts: Number of participants positive for anti-drug antibodies (ADA) to determine incidence of ADA | From Cycle 1 Day 1 through end of treatment or for up to 1 year (Cycles are 21 days or 28 days depending on the assigned dosing schedule)
  Number of participants positive for anti-drug antibodies (ADA) from all participants receiving BT8009 as a monotherapy or in combination with pembrolizumab
Part D: Number of participants with treatment emergent adverse events receiving BT8009 as a monotherapy to assess safety and tolerability in participants with normal renal function or mild renal insufficiency. | From cycle 1 day 1 until at least 30 days after the end of treatment
  Number of participants with advanced solid tumor malignancies associated with Nectin-4 expression receiving BT8009 with normal renal function or mild renal insufficiency who experience treatment-emergent adverse events using CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith McKean, MD, MPH, Study Chair — Tennessee Oncology
Locations (24):
- United States (9):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Ocala Oncology Center, Ocala, Florida
  - Advent Health, Orlando, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Ospedale San Raffaele, Milan
- Spain (5):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - START Madrid Fundacion Jimenez Diaz, Madrid
  - Next Oncology - Hospital Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Marques de Valdecilla, Santander
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Baldini C, Verlingue L, Goldschmidt V, Doger de Speville B, Lostes J, Italiano A, Cousin S, Falchook GS, Necchi A, Reig Torras O, Fontana E, Carter L, Rodon Ahnert J, Brown JR, DeMars LR, Josephs K, Dickson A, Xu C, Bader J, Campbell C, Sharma R, McKean M. First-in-Human, Phase I/II Dose Escalation and Expansion Study of Zelenectide Pevedotin in Patients With Advanced Solid Tumors: Results From Monotherapy Dose Escalation. J Clin Oncol. 2025 Dec 10;43(35):3728-3738. doi: 10.1200/JCO-25-00559. Epub 2025 Nov 6. PMID 41197088
- [Derived] Klumper N, Eckstein M, Holzel M, Herrmann K, Hadaschik B, Grunwald V. Re: First-in-Human Study of the Radioligand 68Ga-N188 Targeting Nectin-4 for PET/CT Imaging of Advanced Urothelial Carcinoma: Navigating Metastatic Urothelial Cancer with Nectin-4 PET/CT. Eur Urol. 2023 Nov;84(5):514-515. doi: 10.1016/j.eururo.2023.05.029. Epub 2023 Jun 5. No abstract available. PMID 37286457